CLINICAL TRIAL: NCT03587714
Title: Prevalence of Hepatitis c Virus Infection Among Rheumatological Patients
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Manal Hassanien, principle investigaror, Assiut University
Other Study IDs: Hepatitis C
Record Dates: First submitted 2018-07-04; First posted 2018-07-16 (Actual); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — Patients' serum samples were screened for the presence of anti-HCV antibodies. All Patients were further evaluated for the presence of HCV ribonucleic acid by reverse transcriptase polymerase chain reaction (RT-PCR)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: HCV RT-PCR — HCV ribonucleic acid by reverse transcriptase polymerase chain reaction (RT-PCR)

SUMMARY:
Egypt has the highest prevalence of hepatitis C virus (HCV) in the world. In 2015, the prevalence of HCV RNA was found to be 7.0%.(1) The prevalence of HCV was studied in Rheumatoid arthritis in few studies(2,3), but to our knowledge, no previous work studied it in other rheumatologic diseases.

DETAILED DESCRIPTION:
Egypt has the highest prevalence of hepatitis C virus (HCV) in the world. In 2015, the prevalence of HCV RNA was found to be 7.0%.(1) The prevalence of HCV was studied in Rheumatoid arthritis in few studies(2,3), but to our knowledge, no previous work studied it in other rheumatologic diseases.

This study aims at detecting the prevalence of subclinical HCV infection in different rheumatologic disease groups in Egypt.

Consecutive patients with different rheumatologic diseases from seven- geographically different- rheumatology departments were prospectively studied. None of the patients was known to have previous HCV infection. Patients' serum samples were screened for the presence of anti-HCV antibodies. Patients with positive serology were further evaluated for the presence of HCV ribonucleic acid by reverse transcriptase polymerase chain reaction (RT-PCR)

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with different rheumatologic diseases from seven- geographically different- rheumatology departments were prospectively studied. None of the patients was known to have previous HCV infection

Exclusion Criteria:

* pregnancy and end organ failure

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All rheumatologic and other muscloskeletal diseased patients attending Rheumatology clinic Assuit university hospital
Sampling Method: Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
HCV RT-PCR | 3 months
  positive

CONTACTS AND LOCATIONS:
Overall Officials: Manal Hassanien, MD, Principal Investigator — Assiut University
Locations (1):
- Assiut governorate, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
detecting the prevalence of subclinical HCV infection in different rheumatologic disease groups in Egypt
Supporting Information: Study Protocol, SAP
Time Frame: 3 months